CLINICAL TRIAL: NCT01594359
Title: Efficacy of Iron Biofortified Beans in Improving the Iron Status of Rwandan Adolescent Girls: A Randomized Control Trial
Brief Title: Nutrition Study of Effect of High Iron Beans on Iron Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: HarvestPlus (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Principle Investigator, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Project #8209
Record Dates: First submitted 2012-05-03; First posted 2012-05-09 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Iron Deficiency
Keywords: Ferritin
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High iron bean (Active Comparator): High-iron bean
  Interventions: Other: Biofortified beans
- Low iron bean (Placebo Comparator): Low-iron bean
  Interventions: Other: BEAN

INTERVENTIONS:
Other: Biofortified beans — Comparison of two types of the common bean that are similar in all aspects except their iron concentration - one has a high iron concentration while the other has low iron concentration
  Arms: High iron bean
Other: BEAN — Placebo
  Arms: Low iron bean

SUMMARY:
The purpose of this study is to determine whether beans bred to have a high iron content are effective in improving the iron status of young women.

DETAILED DESCRIPTION:
The goal of the study is to determine the efficacy of biofortified beans in improving the iron status of young women in Rwanda.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adolescent subjects of reproductive age with low iron stores with or without mild anemia, who are otherwise healthy, will be enrolled in the study

Exclusion Criteria:

* Pregnant, lactating, severe anemia, low BMI would be excluded

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Improved iron status | 1 year
  Improvement in serum ferritin

SECONDARY OUTCOMES:
Improved physical and cognitive performance | 1 year
  Tests on physical performance using accelerometers and breath tests; cognitive tests

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Hurrell, PhD, Principal Investigator — ETH Zurich
Locations (2):
- Rwanda (2):
  - National University of Rwanda, Butare, Kigali
  - Kigali, Kigali

REFERENCES:
- [Derived] Luna SV, Pompano LM, Lung'aho M, Gahutu JB, Haas JD. Increased Iron Status during a Feeding Trial of Iron-Biofortified Beans Increases Physical Work Efficiency in Rwandan Women. J Nutr. 2020 May 1;150(5):1093-1099. doi: 10.1093/jn/nxaa016. PMID 32006009
- [Derived] Wenger MJ, Rhoten SE, Murray-Kolb LE, Scott SP, Boy E, Gahutu JB, Haas JD. Changes in Iron Status Are Related to Changes in Brain Activity and Behavior in Rwandan Female University Students: Results from a Randomized Controlled Efficacy Trial Involving Iron-Biofortified Beans. J Nutr. 2019 Apr 1;149(4):687-697. doi: 10.1093/jn/nxy265. PMID 30926992
- [Derived] Murray-Kolb LE, Wenger MJ, Scott SP, Rhoten SE, Lung'aho MG, Haas JD. Consumption of Iron-Biofortified Beans Positively Affects Cognitive Performance in 18- to 27-Year-Old Rwandan Female College Students in an 18-Week Randomized Controlled Efficacy Trial. J Nutr. 2017 Nov;147(11):2109-2117. doi: 10.3945/jn.117.255356. Epub 2017 Sep 27. PMID 28954841
- [Derived] Haas JD, Luna SV, Lung'aho MG, Wenger MJ, Murray-Kolb LE, Beebe S, Gahutu JB, Egli IM. Consuming Iron Biofortified Beans Increases Iron Status in Rwandan Women after 128 Days in a Randomized Controlled Feeding Trial. J Nutr. 2016 Aug;146(8):1586-92. doi: 10.3945/jn.115.224741. Epub 2016 Jun 29. PMID 27358417